CLINICAL TRIAL: NCT04395352
Title: Effectiveness of EndoCuff Vision in Improving Adenoma Detection Rate in a Large Screening-Related Cohort
Brief Title: Effectiveness of Endocuff Vision in Improving ADR
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: HREBA.CC-19-0257
Record Dates: First submitted 2020-04-28; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Pre-ECV: Patients having undergone colonoscopy prior to the introduction of ECV (November 1 2018 to April 30 2019).
- ECV: Patients having undergone colonoscopy after the introduction of ECV (June 1 2019 to November 30 2019).
  Interventions: Device: Endocuff Vision (ECV)

INTERVENTIONS:
Device: Endocuff Vision (ECV) — Detachable disposable (single-use) device that fits over the distal colonoscope end.
  Groups: ECV

SUMMARY:
The goal of distal attachment devices is to enhance an endoscopist's adenoma detection rate (ADR). A device called EndoCuff Vision (ECV) has been introduced that employs a single row of flexible arms to evert colonic folds, thus optimizing mucosal visualization and enhancing ADR. ECV has been shown to be efficacious in improving ADR within the context of randomized trials. However, no 'real-world' studies have been published assessing the effectiveness of ECV in non-trial settings. The primary objective of this study is to assess the effect of ECV use on ADR in a routine screening-related population.

ELIGIBILITY:
Inclusion Criteria:

adult patients undergoing colonoscopy.

Exclusion Criteria:

* single balloon- or double balloon-assisted colonoscopy;
* planned advanced polypectomy or endoscopic mucosal resection (EMR);
* planned endoscopic post-polypectomy or post-EMR surveillance;
* known active diverticulitis;
* known colonic stricture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing screening-related colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 15816 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate (ADR) | Intra-procedural
  Proportion of an endoscopist's screening-related colonoscopies during which one or more adenoma was biopsied or removed

SECONDARY OUTCOMES:
Adenoma detection rate among patients with positive fecal immunochemical tests | Intra-procedural
  Proportion of an endoscopist's colonoscopies performed for +fecal immunochemical test (FIT), or indications other than positive FIT during which one or more adenoma was biopsied or removed. In order to be included in the non-FIT ADR category, a patient must not have undergone a colonoscopy at CCSC within the last four years of the index procedure.
SSADR (sessile serrated adenoma detection rate) | Intra-procedural
  Proportion of an endoscopist's screening-related colonoscopies during which one or more sessile serrated adenoma was biopsied or removed
CIR (cecal intubation rate) | Intra-procedural
  Proportion of an endoscopist's screening-related procedures in which the cecal pole is intubated, as landmarked by direct visualization of the appendiceal orifice, ileocecal valve, or both.
Procedure time | Intra-procedural
  Total time spent by an endoscopist from the start of the colonoscopy procedure (insertion of the colonoscope through the anus) to the end of the colonoscopy (removal of the colonoscope from the anus). This variable will be calculated only for cases in which no pathology was encountered.
Nurse-assessed patient comfort scores (NAPCOMs) | Intra-procedural
  Validated score for determining patients' procedural comfort. Scored from 0 to 9, with higher scores indicating higher discomfort intensity, frequency, and/or duration.
Number of patients with immediate adverse events | Day 1
  Adverse events occurring at the time of colonoscopy or before discharge, including bleeding or perforation.
Number of patients with delayed adverse events | Within 30 days of index procedure
  Adverse events within 30 days of the index procedure, including delayed bleeding, delayed perforation, or acute healthcare utilization (emergency department visit or hospital admission) for any other reasons deemed related to index colonoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Forzani and MacPhail Colon Cancer Screening Centre (CCSC), Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No